CLINICAL TRIAL: NCT03003052
Title: Assessing Current Clinical Concepts in Dental Practice
Status: Recruiting | Type: Observational
Sponsor: The Campbell Clinic, UK (Industry)
Responsible Party: Sponsor
Other Study IDs: TCC-RD-01
Record Dates: First submitted 2016-12-19; First posted 2016-12-26 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Dental Implant
Keywords: dental implants; edentulous; dental hygiene; evidence-based dentistry
MeSH Terms: conditions — Mouth, Edentulous | interventions — Dental Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Dental implants — Data collection from pre-implant assessment, implant surgery, and hygiene recall appointments, to assess implant survival and success.

SUMMARY:
This purpose of this database is to collect, store and use appropriately derived data from routine patient care in a specialist dental practice. Comprehensive observational data will be gathered, systematically organised and be continuously updated. This data will be used to evaluate treatment outcomes and identify areas for improvement. This will contribute to the existing evidence base to validate new and current clinical concepts in dentistry. Patient consent will be sought for this, and all data extracted from patient notes will be stored and used anonymously. Use of the Oral Health Impact Profile (OHIP) -14 questionnaire pre and post treatment will be used to assess patient satisfaction with outcomes.

DETAILED DESCRIPTION:
Specialist dentistry uses a combination of techniques resulting from joint decisions between clinicians and patients, aimed at giving the patient what is perceived to be the best possible outcome. However, as new techniques and approaches develop, there is capacity for more evidence to justify one treatment option over another, both clinically and most importantly, from the patient perspective.

The aim of this project is to set up a research database which will enable the collection and storage of appropriately derived data from routine patient care and from patient questionnaires (using OHIP-14). This data will be used in cohort studies/case series reports/comparative studies with other practices.

It is believed that this process will provide an effective way of evidencing predictable outcomes, assist in the development of improved clinical techniques, provide additional guidance and support for patients, and further clinical research in dental practice. In addition, implementation of studies to track patient satisfaction with clinical outcomes will provide advanced support in the decision making process.

All adult patients treated at The Campbell Clinic will be approached for consent. This will be an ongoing process, to maximize sample size. Treatment decisions will be continue to be made jointly by clinician and patient and will not be altered by participation in this study. Patient consent will be sought, and all data will be anonymised for storage in the database.

ELIGIBILITY:
Inclusion Criteria:

1. be a patient at The Campbell Clinic
2. be planning to undergo or have undergone specialist dental treatment, usually involved dental implants
3. be able to read and understand Patient Information Sheet
4. Have signed informed consent form

Exclusion Criteria:

1. concern that patient has not understood patient information sheet (e.g. due to language /interpretation issues)
2. not willing to sign consent form
3. any medical condition/medication that might compromise implant success

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients treated at the Campbell Clinic, with focus on dental implants
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-01; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Implant Success - clinical measures | up to 4 years
  Assessment of implant success (signs of implant mucositis peri-implantitis), functionality and aesthetic results. Categorised/grouped by surgery type: single/multiple implant, use of sinus lift, and other variables.

SECONDARY OUTCOMES:
Implant Success - patient defined | up to 4 years
  Assessment of functionality and aesthetic results from patient perspective - measured using OHIP-14 patient questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Campbell, Principal Investigator — The Campbell Clinic
Locations (1):
- The Campbell Clinic, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No